CLINICAL TRIAL: NCT03112031
Title: A Randomized Trial of Tamoxifen Combined With Amphotericin B and Fluconazole for Cryptococcal Meningitis
Brief Title: Treatment With Tamoxifen in Cryptococcal Meningitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Cho Ray Hospital (Other); University of Liverpool (Other); University of Rochester (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28CN
Record Dates: First submitted 2017-03-29; First posted 2017-04-13 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Meningitis Streptococcal; Hiv; Meningitis; Meningoencephalitis
Keywords: Tamoxifen; Cryptococcal meningitis; Cryptococcus neoformans; Human immunodeficiency virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Meningitis; Meningoencephalitis; Meningitis, Cryptococcal; Cryptococcosis | interventions — Tamoxifen; Amphotericin B; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen augmented antifungal therapy (Experimental): Tamoxifen 300mg/day for 2 weeks, combined with standard antifungal therapy (amphotericin B 1mg/kg/day combined with fluconazole 800mg/day for the first 2 weeks followed by fluconazole 800mg/day for 8 weeks)
  Interventions: Drug: Tamoxifen; Drug: Amphotericin B; Drug: Fluconazole
- Standard antifungal therapy (Active Comparator): Amphotericin B 1mg/kg/day combined with fluconazole 800mg/day for the first 2 weeks followed by fluconazole 800mg/day for 8 weeks.
  Interventions: Drug: Amphotericin B; Drug: Fluconazole

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen will be given orally in a dose of 300mg/day for the first 14 days following randomization. It will be administered by nasogastric tube where patients are unconscious. The Tamoxifen will be administered in the morning combined with amphotericin and fluconazole dose.
  Other Names: Nolvadex - D
  Arms: Tamoxifen augmented antifungal therapy
Drug: Amphotericin B — Patients will receive amphotericin 1mg/kg/day i.v. once daily orally for the first 2 weeks.
  Other Names: Amphotret
Drug: Fluconazole — Patients will receive fluconazole 800mg once daily orally for the first 2 weeks. Amphotericin and fluconazole will be administered simultaneously. After the first 2 weeks of study treatment, all patients will receive fluconazole 800mg/day for 8 further weeks, until the study end.
  Other Names: Zolmed 200

SUMMARY:
The purpose of this study is to develop initial efficacy, feasibility, and safety data regarding the use of Tamoxifen in combination with amphotericin B and fluconazole in the treatment of cryptococcal meningitis. The results of the study will inform the design and feasibility of a larger study powered to a survival endpoint. The study hypothesis is that adding tamoxifen to standard antifungal therapy increases the rate of clearance of yeast from cerebrospinal fluid. Increased rates of clearance of yeast from cerebrospinal fluid have previously been associated with improved clinical outcomes, including survival and disability.

DETAILED DESCRIPTION:
A randomized, open-label trial with 2 parallel arms: standard antifungal therapy versus tamoxifen augmented antifungal therapy during the first 2 weeks (induction phase) of treatment. The study will recruit in two sites in Ho Chi Minh City: the Hospital for Tropical Diseases (HTD), and Cho Ray Hospital (CRH). 25 patients will be enrolled into the two study arms (intervention versus control). All anti-fungal administration will be directly observed by ward staff.

Intervention arm: Induction phase treatment (days 1-14): Tamoxifen will be given orally in a dose of 300mg/day for the first 14 days following randomization. It will be administered by nasogastric tube where patients are unconscious. In addition patients will receive amphotericin 1mg/kg once daily iv and fluconazole 800mg once daily orally. The tamoxifen will be administered in the morning combined with amphotericin and fluconazole dose.

Control arm: Induction phase treatment (days 1-14): Patients will receive amphotericin 1mg/kg/day combined with fluconazole 800mg once daily for the first 2 weeks. Amphotericin and fluconazole will be administered simultaneously.

The primary efficacy endpoint will be the rate of clearance of yeast cells from cerebrospinal fluid (CSF) over the first 2 weeks following randomisation. Patients will be followed for 10 weeks, which is conventional in clinical trials in cryptococcal meningitis. After the first 2 weeks of study treatment, all patients will receive fluconazole 800mg/day for 8 further weeks, until the study end. At this point, HIV infected patients will be switched to long term secondary prophylaxis with fluconazole 200mg/day as per standard practice. For HIV uninfected patients, the decision to continue antifungal treatment, and at which dose, will be made on a case by case basis by the attending physician in consultation with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cryptococcal meningitis (CM) defined as a syndrome consistent with CM and one or more of:

  * positive CSF India ink (budding encapsulated yeasts),
  * C. neoformans cultured from CSF or blood,
  * positive cryptococcal antigen Lateral Flow Antigen Test (LFA) in CSF
* Informed consent to participate given by patient or acceptable representative
* Known HIV infection status, or patient agrees to HIV testing on this admission

Exclusion Criteria:

* Pregnancy or breast-feeding
* History of thromboembolic disease such as pulmonary embolism or deep venous thrombosis
* On anti-coagulant medication
* On medication known to prolong the QT interval other than fluconazole, such as fluoroquinolones or antidepressants.
* Known cardiac conduction defect including long QT syndromes
* QTc at baseline > 500ms
* Currently receiving treatment for cryptococcal meningitis and having received > 4 days of anti-cryptococcal meningitis therapy
* Known allergy to Tamoxifen
* Currently or history of receiving treatment with Tamoxifen for breast cancer or other indication
* Current or history of uterine cancer including endometrial cancer and uterine sarcoma
* Renal failure (defined as creatinine >3*ULN (upper limit of normal), despite adequate hydration)
* Failure to consent - the patient, or if they are incapacitated, their responsible relative, declines to enter the study
* Allergy to amphotericin B or fluconazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Early Fungicidal Activity (EFA), i.e. the rate of clearance of yeast from cerebrospinal fluid | over the first 2 weeks following randomisation
  In the trial, lumbar punctures are scheduled on days 1, 3, 7, 14, and additionally as clinically indicated. Whenever a lumbar puncture is performed, the study team will determine the amount of viable yeast in CSF through culture. Based on the patients' longitudinal quantitative yeast count measurements, EFA will be determined as previously described e.g. see N Engl J Med 2016; 374:542-54

SECONDARY OUTCOMES:
Survival until 10 weeks after randomization | 10 weeks after randomisation
  International treatment guidelines recommend 10 weeks of high dose antifungal therapy for cryptococcal meningitis - an initial phase of amphotericin based induction therapy for 2 weeks followed by 8 weeks of moderate to high dose fluconazole. The rate of survival until this 10 week period of therapy is completed is a frequent endpoint in trials of treatment for cryptococcal meningitis.
Disability at 10 weeks | at 10 weeks
  Disability is an expected consequence of cryptococcal meningitis, including blindness, deafness and other focal neurological deficits. Neurological disability will be assessed using the modified Rankin score and the Two Simple Questions, and the results of each test combined and classified as good, intermediate, severe disability, or death, as we have previously published.
Adverse events | During hospital stay, an average of 10 weeks
  The proportion of patients with any grade 3 or 4 adverse event, serious adverse event, or unexpected serious adverse event will be compared between treatment groups.
Rate of IRIS until 10 weeks (in HIV infected patients only) | until 10 weeks
  The investigators will model the rate of IRIS over time with a cause-specific hazards model taking into account the competing risk of prior death.
Rate of Cryptococcal meningitis relapse | until 10 weeks
  A pragmatic definition of relapse will be used. This is defined as either intensification of antifungal therapy above that according to the study antifungal schedule, or readmission for treatment of cryptococcal disease.
QT prolongation | During hospital stay, an average of 10 weeks
  Prolongation of the QT interval is a potential side-effect of both Tamoxifen and fluconazole, although it is not clear that either drug increases the risk of Torsade de Pointes, a potentially life-threatening arrhythmia. The QT interval will be estimated manually from 3 chest and 3 limb leads from a high resolution (50mm/sec) 12-lead ECG. The median value will be determined and used to calculate the corrected QT interval (QTc) using using Framingham's formula
Visual deficit at 10 weeks | at 10 weeks
  Visual deficit occurs in 5-40% of patients with cryptococcal meningitis depending upon underlying immune status. The pathogenesis is unclear. The study team will compare the incidence of blindness and other visual deficit between treatment groups. Visual deficit will be assessed using a simple 6 point scale.
Time to new neurological event or death until 10 weeks | until 10 weeks
  A neurological event is defined as a fall in Glasgow coma score by ≥2 points for ≥2 days from the highest previously recorded Glasgow coma score (including baseline) or the occurrence of any of the following adverse events: cerebellar symptoms, coma, hemiplegia, paraplegia, seizures, cerebral herniation, new onset blindness or deafness, or cranial nerve palsy.
Longitudinal measurements of intracranial pressure during the first 2 weeks | during the first 2 weeks
  Intracranial pressure (ICP) will be measured at study entry, day 3, 7, and 14, and at other times as clinically indicated. The decline in raised intracranial pressure over the first 2 weeks will be modelled and compared between treatment arms.
CD4 count at 10 weeks | at 10 weeks
  CD4 count measurement is indicated in HIV infected patients, and CD4 lymphopenia has been described in HIV uninfected patients with cryptococcal meningitis. Moreover, Tamoxifen may reduce CD4 cell apoptosis which may be beneficial.
Blood and CSF concentrations of amphotericin, Tamoxifen and fluconazole | During hospital stay, an average of 10 weeks
  All patients will undergo pharmacokinetic sampling to enable the description of the concentrations of Tamoxifen and fluconazole in plasma and CSF, and of amphotericin in blood, and relate these to the rate of clearance of yeast from CSF.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Day, MD, Principal Investigator — Oxford University Clinical Research Unit
Locations (3):
- Vietnam (3):
  - Cho Ray Hospital, Ho Chi Minh City
  - Hospital for Tropical Diseases, Ho Chi Minh City
  - Oxford University Clinical Research Unit, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park BJ, Wannemuehler KA, Marston BJ, Govender N, Pappas PG, Chiller TM. Estimation of the current global burden of cryptococcal meningitis among persons living with HIV/AIDS. AIDS. 2009 Feb 20;23(4):525-30. doi: 10.1097/QAD.0b013e328322ffac. PMID 19182676
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Chen S, Sorrell T, Nimmo G, Speed B, Currie B, Ellis D, Marriott D, Pfeiffer T, Parr D, Byth K. Epidemiology and host- and variety-dependent characteristics of infection due to Cryptococcus neoformans in Australia and New Zealand. Australasian Cryptococcal Study Group. Clin Infect Dis. 2000 Aug;31(2):499-508. doi: 10.1086/313992. Epub 2000 Sep 7. PMID 10987712
- [Background] Chau TT, Mai NH, Phu NH, Nghia HD, Chuong LV, Sinh DX, Duong VA, Diep PT, Campbell JI, Baker S, Hien TT, Lalloo DG, Farrar JJ, Day JN. A prospective descriptive study of cryptococcal meningitis in HIV uninfected patients in Vietnam - high prevalence of Cryptococcus neoformans var grubii in the absence of underlying disease. BMC Infect Dis. 2010 Jul 9;10:199. doi: 10.1186/1471-2334-10-199. PMID 20618932
- [Background] Perfect JR, Dismukes WE, Dromer F, Goldman DL, Graybill JR, Hamill RJ, Harrison TS, Larsen RA, Lortholary O, Nguyen MH, Pappas PG, Powderly WG, Singh N, Sobel JD, Sorrell TC. Clinical practice guidelines for the management of cryptococcal disease: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2010 Feb 1;50(3):291-322. doi: 10.1086/649858. PMID 20047480
- [Background] Day JN, Chau TTH, Wolbers M, Mai PP, Dung NT, Mai NH, Phu NH, Nghia HD, Phong ND, Thai CQ, Thai LH, Chuong LV, Sinh DX, Duong VA, Hoang TN, Diep PT, Campbell JI, Sieu TPM, Baker SG, Chau NVV, Hien TT, Lalloo DG, Farrar JJ. Combination antifungal therapy for cryptococcal meningitis. N Engl J Med. 2013 Apr 4;368(14):1291-1302. doi: 10.1056/NEJMoa1110404. PMID 23550668
- [Background] Beardsley J, Wolbers M, Kibengo FM, Ggayi AB, Kamali A, Cuc NT, Binh TQ, Chau NV, Farrar J, Merson L, Phuong L, Thwaites G, Van Kinh N, Thuy PT, Chierakul W, Siriboon S, Thiansukhon E, Onsanit S, Supphamongkholchaikul W, Chan AK, Heyderman R, Mwinjiwa E, van Oosterhout JJ, Imran D, Basri H, Mayxay M, Dance D, Phimmasone P, Rattanavong S, Lalloo DG, Day JN; CryptoDex Investigators. Adjunctive Dexamethasone in HIV-Associated Cryptococcal Meningitis. N Engl J Med. 2016 Feb 11;374(6):542-54. doi: 10.1056/NEJMoa1509024. PMID 26863355
- [Background] Loyse A, Dromer F, Day J, Lortholary O, Harrison TS. Flucytosine and cryptococcosis: time to urgently address the worldwide accessibility of a 50-year-old antifungal. J Antimicrob Chemother. 2013 Nov;68(11):2435-44. doi: 10.1093/jac/dkt221. Epub 2013 Jun 20. PMID 23788479
- [Background] Butts A, Koselny K, Chabrier-Rosello Y, Semighini CP, Brown JC, Wang X, Annadurai S, DiDone L, Tabroff J, Childers WE Jr, Abou-Gharbia M, Wellington M, Cardenas ME, Madhani HD, Heitman J, Krysan DJ. Estrogen receptor antagonists are anti-cryptococcal agents that directly bind EF hand proteins and synergize with fluconazole in vivo. mBio. 2014 Feb 11;5(1):e00765-13. doi: 10.1128/mBio.00765-13. PMID 24520056
- [Background] Perez EA, Gandara DR, Edelman MJ, O'Donnell R, Lauder IJ, DeGregorio M. Phase I trial of high-dose tamoxifen in combination with cisplatin in patients with lung cancer and other advanced malignancies. Cancer Invest. 2003;21(1):1-6. doi: 10.1081/cnv-120016397. PMID 12643003
- [Background] Bergan RC, Reed E, Myers CE, Headlee D, Brawley O, Cho HK, Figg WD, Tompkins A, Linehan WM, Kohler D, Steinberg SM, Blagosklonny MV. A Phase II study of high-dose tamoxifen in patients with hormone-refractory prostate cancer. Clin Cancer Res. 1999 Sep;5(9):2366-73. PMID 10499606
- [Background] Ducharme J, Fried K, Shenouda G, Leyland-Jones B, Wainer IW. Tamoxifen metabolic patterns within a glioma patient population treated with high-dose tamoxifen. Br J Clin Pharmacol. 1997 Feb;43(2):189-93. doi: 10.1046/j.1365-2125.1997.05029.x. PMID 9131952
- [Background] Smith DC, Trump DL. A phase I trial of high-dose oral tamoxifen and CHOPE. Cancer Chemother Pharmacol. 1995;36(1):65-8. doi: 10.1007/BF00685734. PMID 7720178
- [Background] Trump DL, Smith DC, Ellis PG, Rogers MP, Schold SC, Winer EP, Panella TJ, Jordan VC, Fine RL. High-dose oral tamoxifen, a potential multidrug-resistance-reversal agent: phase I trial in combination with vinblastine. J Natl Cancer Inst. 1992 Dec 2;84(23):1811-6. doi: 10.1093/jnci/84.23.1811. PMID 1359155
- [Background] Wiseman H, Cannon M, Arnstein HR. Observation and significance of growth inhibition of Saccharomyces cerevisiae (A224A) by the anti-oestrogen drug tamoxifen. Biochem Soc Trans. 1989 Dec;17(6):1038-9. doi: 10.1042/bst0171038. No abstract available. PMID 2697611
- [Background] Beggs WH. Anti-Candida activity of the anti-cancer drug tamoxifen. Res Commun Chem Pathol Pharmacol. 1993 Apr;80(1):125-8. PMID 8488339
- [Background] Beggs WH. Comparative activities of miconazole and the anticancer drug tamoxifen against Candida albicans. J Antimicrob Chemother. 1994 Jul;34(1):186-7. doi: 10.1093/jac/34.1.186. No abstract available. PMID 7961210
- [Background] Dolan K, Montgomery S, Buchheit B, Didone L, Wellington M, Krysan DJ. Antifungal activity of tamoxifen: in vitro and in vivo activities and mechanistic characterization. Antimicrob Agents Chemother. 2009 Aug;53(8):3337-46. doi: 10.1128/AAC.01564-08. Epub 2009 Jun 1. PMID 19487443
- [Background] Spitzer M, Griffiths E, Blakely KM, Wildenhain J, Ejim L, Rossi L, De Pascale G, Curak J, Brown E, Tyers M, Wright GD. Cross-species discovery of syncretic drug combinations that potentiate the antifungal fluconazole. Mol Syst Biol. 2011 Jun 21;7:499. doi: 10.1038/msb.2011.31. PMID 21694716
- [Background] Lien EA, Solheim E, Ueland PM. Distribution of tamoxifen and its metabolites in rat and human tissues during steady-state treatment. Cancer Res. 1991 Sep 15;51(18):4837-44. PMID 1893376
- [Background] Lien EA, Wester K, Lonning PE, Solheim E, Ueland PM. Distribution of tamoxifen and metabolites into brain tissue and brain metastases in breast cancer patients. Br J Cancer. 1991 Apr;63(4):641-5. doi: 10.1038/bjc.1991.147. PMID 2021551
- [Background] Senkus E, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rutgers E, Zackrisson S, Cardoso F; ESMO Guidelines Committee. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v8-30. doi: 10.1093/annonc/mdv298. No abstract available. PMID 26314782
- [Background] Tormey DC, Lippman ME, Edwards BK, Cassidy JG. Evaluation of tamoxifen doses with and without fluoxymesterone in advanced breast cancer. Ann Intern Med. 1983 Feb;98(2):139-44. doi: 10.7326/0003-4819-98-2-139. PMID 6824247
- [Background] Muanza T, Shenouda G, Souhami L, Leblanc R, Mohr G, Corns R, Langleben A. High dose tamoxifen and radiotherapy in patients with glioblastoma multiforme: a phase IB study. Can J Neurol Sci. 2000 Nov;27(4):302-6. doi: 10.1017/s0317167100001049. PMID 11097520
- [Background] Skapek SX, Anderson JR, Hill DA, Henry D, Spunt SL, Meyer W, Kao S, Hoffer FA, Grier HE, Hawkins DS, Raney RB. Safety and efficacy of high-dose tamoxifen and sulindac for desmoid tumor in children: results of a Children's Oncology Group (COG) phase II study. Pediatr Blood Cancer. 2013 Jul;60(7):1108-12. doi: 10.1002/pbc.24457. Epub 2012 Dec 31. PMID 23281268
- [Background] Powles TJ, Ashley S, Tidy A, Smith IE, Dowsett M. Twenty-year follow-up of the Royal Marsden randomized, double-blinded tamoxifen breast cancer prevention trial. J Natl Cancer Inst. 2007 Feb 21;99(4):283-90. doi: 10.1093/jnci/djk050. PMID 17312305
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Pollack IF, DaRosso RC, Robertson PL, Jakacki RL, Mirro JR Jr, Blatt J, Nicholson S, Packer RJ, Allen JC, Cisneros A, Jordan VC. A phase I study of high-dose tamoxifen for the treatment of refractory malignant gliomas of childhood. Clin Cancer Res. 1997 Jul;3(7):1109-15. PMID 9815790
- [Background] Drew BJ, Ackerman MJ, Funk M, Gibler WB, Kligfield P, Menon V, Philippides GJ, Roden DM, Zareba W; American Heart Association Acute Cardiac Care Committee of the Council on Clinical Cardiology, the Council on Cardiovascular Nursing, and the American College of Cardiology Foundation. Prevention of torsade de pointes in hospital settings: a scientific statement from the American Heart Association and the American College of Cardiology Foundation. Circulation. 2010 Mar 2;121(8):1047-60. doi: 10.1161/CIRCULATIONAHA.109.192704. Epub 2010 Feb 8. No abstract available. PMID 20142454
- [Background] Hamlin RL. A search to predict potential for drug-induced cardiovascular toxicity. Toxicol Pathol. 2006;34(1):75-80. doi: 10.1080/01926230500419439. PMID 16507547
- [Background] Johannesen L, Vicente J, Mason JW, Sanabria C, Waite-Labott K, Hong M, Guo P, Lin J, Sorensen JS, Galeotti L, Florian J, Ugander M, Stockbridge N, Strauss DG. Differentiating drug-induced multichannel block on the electrocardiogram: randomized study of dofetilide, quinidine, ranolazine, and verapamil. Clin Pharmacol Ther. 2014 Nov;96(5):549-58. doi: 10.1038/clpt.2014.155. Epub 2014 Jul 23. PMID 25054430
- [Background] Liu XK, Katchman A, Ebert SN, Woosley RL. The antiestrogen tamoxifen blocks the delayed rectifier potassium current, IKr, in rabbit ventricular myocytes. J Pharmacol Exp Ther. 1998 Dec;287(3):877-83. PMID 9864267
- [Background] Asp ML, Martindale JJ, Metzger JM. Direct, differential effects of tamoxifen, 4-hydroxytamoxifen, and raloxifene on cardiac myocyte contractility and calcium handling. PLoS One. 2013 Oct 24;8(10):e78768. doi: 10.1371/journal.pone.0078768. eCollection 2013. PMID 24205315
- [Background] He J, Kargacin ME, Kargacin GJ, Ward CA. Tamoxifen inhibits Na+ and K+ currents in rat ventricular myocytes. Am J Physiol Heart Circ Physiol. 2003 Aug;285(2):H661-8. doi: 10.1152/ajpheart.00686.2002. Epub 2003 Apr 17. PMID 12702490
- [Background] Han S, Zhang Y, Chen Q, Duan Y, Zheng T, Hu X, Zhang Z, Zhang L. Fluconazole inhibits hERG K(+) channel by direct block and disruption of protein trafficking. Eur J Pharmacol. 2011 Jan 10;650(1):138-44. doi: 10.1016/j.ejphar.2010.10.010. Epub 2010 Oct 15. PMID 20951697
- [Background] McMahon JH, Grayson ML. Torsades de pointes in a patient receiving fluconazole for cerebral cryptococcosis. Am J Health Syst Pharm. 2008 Apr 1;65(7):619-23. doi: 10.2146/ajhp070203. PMID 18359968
- [Background] Tatetsu H, Asou N, Nakamura M, Hanaoka N, Matsuno F, Horikawa K, Mitsuya H. Torsades de pointes upon fluconazole administration in a patient with acute myeloblastic leukemia. Am J Hematol. 2006 May;81(5):366-9. doi: 10.1002/ajh.20557. PMID 16628725
- [Background] Frommeyer G, Eckardt L. Drug-induced proarrhythmia: risk factors and electrophysiological mechanisms. Nat Rev Cardiol. 2016 Jan;13(1):36-47. doi: 10.1038/nrcardio.2015.110. Epub 2015 Jul 21. PMID 26194552
- [Background] Zeuli JD, Wilson JW, Estes LL. Effect of combined fluoroquinolone and azole use on QT prolongation in hematology patients. Antimicrob Agents Chemother. 2013 Mar;57(3):1121-7. doi: 10.1128/AAC.00958-12. Epub 2012 Dec 10. PMID 23229485
- [Background] Isbister GK. How do we assess whether the QT interval is abnormal: myths, formulae and fixed opinion. Clin Toxicol (Phila). 2015 May;53(4):189-91. doi: 10.3109/15563650.2015.1014044. Epub 2015 Feb 19. No abstract available. PMID 25695875
- [Background] van der Horst CM, Saag MS, Cloud GA, Hamill RJ, Graybill JR, Sobel JD, Johnson PC, Tuazon CU, Kerkering T, Moskovitz BL, Powderly WG, Dismukes WE. Treatment of cryptococcal meningitis associated with the acquired immunodeficiency syndrome. National Institute of Allergy and Infectious Diseases Mycoses Study Group and AIDS Clinical Trials Group. N Engl J Med. 1997 Jul 3;337(1):15-21. doi: 10.1056/NEJM199707033370103. PMID 9203426
- [Background] Thwaites GE, Nguyen DB, Nguyen HD, Hoang TQ, Do TT, Nguyen TC, Nguyen QH, Nguyen TT, Nguyen NH, Nguyen TN, Nguyen NL, Nguyen HD, Vu NT, Cao HH, Tran TH, Pham PM, Nguyen TD, Stepniewska K, White NJ, Tran TH, Farrar JJ. Dexamethasone for the treatment of tuberculous meningitis in adolescents and adults. N Engl J Med. 2004 Oct 21;351(17):1741-51. doi: 10.1056/NEJMoa040573. PMID 15496623
- [Background] Haddow LJ, Colebunders R, Meintjes G, Lawn SD, Elliott JH, Manabe YC, Bohjanen PR, Sungkanuparph S, Easterbrook PJ, French MA, Boulware DR; International Network for the Study of HIV-associated IRIS (INSHI). Cryptococcal immune reconstitution inflammatory syndrome in HIV-1-infected individuals: proposed clinical case definitions. Lancet Infect Dis. 2010 Nov;10(11):791-802. doi: 10.1016/S1473-3099(10)70170-5. PMID 21029993
- [Background] Pan G, Zhou T, Radding W, Saag MS, Mountz JD, McDonald JM. Calmodulin antagonists inhibit apoptosis of CD4+ T-cells from patients with AIDS. Immunopharmacology. 1998 Aug;40(2):91-103. doi: 10.1016/s0162-3109(98)00018-6. PMID 9826024
- [Background] Brammer KW, Farrow PR, Faulkner JK. Pharmacokinetics and tissue penetration of fluconazole in humans. Rev Infect Dis. 1990 Mar-Apr;12 Suppl 3:S318-26. doi: 10.1093/clinids/12.supplement_3.s318. PMID 2184510
- [Background] Manosuthi W, Chetchotisakd P, Nolen TL, Wallace D, Sungkanuparph S, Anekthananon T, Supparatpinyo K, Pappas PG, Larsen RA, Filler SG, Andes D; BAMSG 3-01 Study Team. Monitoring and impact of fluconazole serum and cerebrospinal fluid concentration in HIV-associated cryptococcal meningitis-infected patients. HIV Med. 2010 Apr;11(4):276-81. doi: 10.1111/j.1468-1293.2009.00778.x. Epub 2009 Dec 8. PMID 20002501
- [Background] Menichetti F, Fiorio M, Tosti A, Gatti G, Bruna Pasticci M, Miletich F, Marroni M, Bassetti D, Pauluzzi S. High-dose fluconazole therapy for cryptococcal meningitis in patients with AIDS. Clin Infect Dis. 1996 May;22(5):838-40. doi: 10.1093/clinids/22.5.838. PMID 8722942
- [Background] Gupta G, Fries BC. Variability of phenotypic traits in Cryptococcus varieties and species and the resulting implications for pathogenesis. Future Microbiol. 2010 May;5(5):775-87. doi: 10.2217/fmb.10.44. PMID 20441549
- [Background] Liu OW, Chun CD, Chow ED, Chen C, Madhani HD, Noble SM. Systematic genetic analysis of virulence in the human fungal pathogen Cryptococcus neoformans. Cell. 2008 Oct 3;135(1):174-88. doi: 10.1016/j.cell.2008.07.046. PMID 18854164
- [Background] Ma H, Hagen F, Stekel DJ, Johnston SA, Sionov E, Falk R, Polacheck I, Boekhout T, May RC. The fatal fungal outbreak on Vancouver Island is characterized by enhanced intracellular parasitism driven by mitochondrial regulation. Proc Natl Acad Sci U S A. 2009 Aug 4;106(31):12980-5. doi: 10.1073/pnas.0902963106. Epub 2009 Jul 27. PMID 19651610
- [Background] Idnurm A, Reedy JL, Nussbaum JC, Heitman J. Cryptococcus neoformans virulence gene discovery through insertional mutagenesis. Eukaryot Cell. 2004 Apr;3(2):420-9. doi: 10.1128/EC.3.2.420-429.2004. PMID 15075272
- [Background] Nelson RT, Hua J, Pryor B, Lodge JK. Identification of virulence mutants of the fungal pathogen Cryptococcus neoformans using signature-tagged mutagenesis. Genetics. 2001 Mar;157(3):935-47. doi: 10.1093/genetics/157.3.935. PMID 11238384
- [Background] Day JN, Hoang TN, Duong AV, Hong CT, Diep PT, Campbell JI, Sieu TP, Hien TT, Bui T, Boni MF, Lalloo DG, Carter D, Baker S, Farrar JJ. Most cases of cryptococcal meningitis in HIV-uninfected patients in Vietnam are due to a distinct amplified fragment length polymorphism-defined cluster of Cryptococcus neoformans var. grubii VN1. J Clin Microbiol. 2011 Feb;49(2):658-64. doi: 10.1128/JCM.01985-10. Epub 2010 Dec 15. PMID 21159929
- [Background] Rapid Advice: Diagnosis, Prevention and Management of Cryptococcal Disease in HIV-Infected Adults, Adolescents and Children. Geneva: World Health Organization; 2011 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK299520/ PMID 26110194
- [Background] Morello KC, Wurz GT, DeGregorio MW. Pharmacokinetics of selective estrogen receptor modulators. Clin Pharmacokinet. 2003;42(4):361-72. doi: 10.2165/00003088-200342040-00004. PMID 12648026
- [Derived] Ngan NTT, Thanh Hoang Le N, Vi Vi NN, Van NTT, Mai NTH, Van Anh D, Trieu PH, Lan NPH, Phu NH, Chau NVV, Lalloo DG, Hope W, Beardsley J, White NJ, Geskus R, Thwaites GE, Krysan D, Tai LTH, Kestelyn E, Binh TQ, Hung LQ, Tung NLN, Day JN. An open label randomized controlled trial of tamoxifen combined with amphotericin B and fluconazole for cryptococcal meningitis. Elife. 2021 Sep 28;10:e68929. doi: 10.7554/eLife.68929. PMID 34581270
- [Derived] Ngan NTT, Mai NTH, Tung NLN, Lan NPH, Tai LTH, Phu NH, Chau NVV, Binh TQ, Hung LQ, Beardsley J, White N, Lalloo D, Krysan D, Hope W, Geskus R, Wolbers M, Nhat LTH, Thwaites G, Kestelyn E, Day J. A randomized open label trial of tamoxifen combined with amphotericin B and fluconazole for cryptococcal meningitis. Wellcome Open Res. 2019 Jan 22;4:8. doi: 10.12688/wellcomeopenres.15010.1. eCollection 2019. PMID 30801037